CLINICAL TRIAL: NCT04205877
Title: The United States Patent Ductus Arteriosus Registry
Brief Title: The U.S. PDA Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Shyam K. Sathanandam, MD, Associate Professor of Pediatrics, University of Tennessee. Director of Cath Lab, Le Bonheur Children's Hospital., Le Bonheur Children's Hospital
Other Study IDs: The U.S. PDA Registry
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Ductus Arteriosus, Patent
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Registry Group: All participants will have the same data collected at the same time points.
  Interventions: Device: Transcatheter PDA Closure

INTERVENTIONS:
Device: Transcatheter PDA Closure — Device utilized for closure of PDA, study is to help assure continued safety and effectiveness of FDA approved Amplatzer Piccolo Occluder device as well as other devices used off label for PDA closure in premature infants less than 2 kg at the time of device implant.

SUMMARY:
The objective of this study is to demonstrate the continued safety and efficacy in a real-world setting of transcatheter device closure of the PDA in premature infants less than 2kg in weight at the time of device implant using the Amplatzer Piccolo Occluder device and other devices performed in the USA.

DETAILED DESCRIPTION:
Based on the IMPACT registry, there are over 6000 transcatheter device closures of PDA that occurs in the United States annually. However, there are no comprehensive data collection tools for this procedure. The current databases do not include multiple data points, or follow-up data, or a section for specific adverse events to be documented. Moreover, until now, there has been no approved devices for PDA closure in children < 2kg. This clinical study is the first of its kind to collect data from all transcatheter device closure of PDA in children < 2kg performed in the USA.This study will be limited to children between 700 to 2000 grams who are the most vulnerable population undergoing this procedure. This will allow us to understand the real world experience (efficacy and safety) of using the Amplatzer Piccolo Occluder and other devices in an extremely vulnerable, yet highly underserved population. The study will allow for standardization of this procedure throughout the country for the small children (<2 kg) with a PDA. This is a multi-center, single arm, observational data collection study. This will be a large population study to help analyze outcomes in subjects <2 kg. The trial has two primary endpoints for safety and effectiveness without formal hypothesis. The safety and effectiveness results will be compared with data reported in the ADO II AS IDE and Continued Access Protocol studies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PDA.
2. Clinical indication for transcatheter PDA closure (discretion of the physician).
3. Weight <2 kg at the time of device implant.

Exclusion Criteria:

1. Weight <700 gm or greater than or equal to 2 kg at the time of device implant.
2. Age < 3 days at the time of device implant.
3. Pre-existing coarctation of the aorta.
4. Pre-existing left pulmonary artery stenosis.
5. Cardiac output that is dependent on right to left shunt through the PDA due to pulmonary hypertension.
6. Intracardiac thrombus that interferes with device implant.
7. Active infection requiring treatment at the time of impant.

Ages: 3 Days to 1 Year | Sex: All
Age Groups: Child
Study Population: The study population is patients with diagnosis of PDA with clinical indication for transcatheter PDA closure, and weigh less than 2 kg at the time of device implant.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular Access Complications (Safety) | 6 months
  Access vessel complications include femoral arterial or femoral/jugular venous complications noted during the procedure, immediately after the procedure or delayed (>24 hours). They range from bleeding from access sites, arterial or venous thrombosis with or without the need for treatment to loss of limb secondary to arterial occlusion.
Valvular Injury (Safety) | 6 months
  Valvular injury includes damage to the tricuspid valve or other cardiac valve resulting in immediate post-procedural valvular dysfunction.
Device Embolization (Safety) | 6 months
  Device embolization includes malposition of the device either during or after the procedure or delayed (>24 hours). The outcome of device embolization ranges from observation, transcatheter retrieval at time of procedure or at a separate time, surgical retrieval, other end organ damage, to mortality.
Pulmonary or Aortic Vessel Stenosis (Safety) | 6 months
  Adjacent vessel stenosis includes a narrowing of the aorta or the left pulmonary artery directly as a consequence of device implantation for PDA closure. Vessel stenosis could happen either during or after the procedure or delayed (>24 hours). The outcome of vessel stenosis ranges from no intervention needed to repeated transcatheter and surgical therapies.
Rate of Effective PDA Closure (Effectiveness) | 6 months
  The effectiveness endpoint is the rate of effective closure of the PDA using a transcatheter device within six months post procedure. If more than one attempt is required, or multiple devices are required during the same procedure, it is still considered effective if there is Grade 0 or Grade 1 shunt, as defined below, at follow-up by transthoracic echocardiography or if a second procedure is not required following the initial attempt. If there is device embolization, adjacent vessel stenosis that required retrieval of the device and replacement during the same procedure with less than Grade 1 shunt during follow-up, it is still considered effective. Conversely, if an AE is noted after the procedure that requires a second procedure for treatment that results in greater than Grade 1 shunt, then the procedure is considered not effective, even if the initial attempt was effective. See protocol for PDA shunt definitions.

SECONDARY OUTCOMES:
Significant obstruction of the left pulmonary artery | 6 months
  Significant obstruction of the left pulmonary artery is defined as less than 30% flow to the left lung by lung perfusion scan or a peak instantaneous gradient in left pulmonary artery
  ≥35 mmHg by echocardiogram if lung perfusion scan is not available or as determined by the interventional cardiologist based on angiographic appearance.
Significant obstruction of the aorta | 6 months
  Significant obstruction of the aorta is defined as a gradient of ≥20 mmHg in the aortic isthmus by invasive aortic catheterization or a mean gradient ≥20 mmHg in the aortic isthmus by echocardiogram if invasive aortic catheterization is not available.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sathanandam, MD, Principal Investigator — National Principal Investigator
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
A Data Management Plan (DMP) will describe procedures used for data review, database cleaning, and issuing and resolving data queries. If appropriate, the DMP may be updated throughout the clinical investigation duration. All revisions will be tracked and document controlled. Subject data will be captured in a validated electronic data capture (EDC) system. Only authorized site personnel will be permitted to enter the CRF data through the EDC system. An electronic audit trail will be used to track any subsequent changes of the entered data.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available when it is collected and added to the national database. It will be available for 12 years.
Access Criteria: Investigators will submit proposal to request data to the Proposal Review Committee. If approved, de-identified data will be shared.

REFERENCES:
- [Result] Tashiro J, Perez EA, Sola JE. Reduced Hospital Mortality With Surgical Ligation of Patent Ductus Arteriosus in Premature, Extremely Low Birth Weight Infants: A Propensity Score-matched Outcome Study. Ann Surg. 2016 Mar;263(3):608-14. doi: 10.1097/SLA.0000000000001228. PMID 25822689
- [Result] Schneider DJ. The patent ductus arteriosus in term infants, children, and adults. Semin Perinatol. 2012 Apr;36(2):146-53. doi: 10.1053/j.semperi.2011.09.025. PMID 22414886
- [Result] Mahoney LT, Coryell KG, Lauer RM. The newborn transitional circulation: a two-dimensional Doppler echocardiographic study. J Am Coll Cardiol. 1985 Sep;6(3):623-9. doi: 10.1016/s0735-1097(85)80123-6. PMID 4031274
- [Result] Philip R, Waller BR 3rd, Agrawal V, Wright D, Arevalo A, Zurakowski D, Sathanandam S. Morphologic characterization of the patent ductus arteriosus in the premature infant and the choice of transcatheter occlusion device. Catheter Cardiovasc Interv. 2016 Feb 1;87(2):310-7. doi: 10.1002/ccd.26287. Epub 2015 Nov 3. PMID 26525611
- [Result] Krichenko A, Benson LN, Burrows P, Moes CA, McLaughlin P, Freedom RM. Angiographic classification of the isolated, persistently patent ductus arteriosus and implications for percutaneous catheter occlusion. Am J Cardiol. 1989 Apr 1;63(12):877-80. doi: 10.1016/0002-9149(89)90064-7. No abstract available. PMID 2929450
- [Result] Pass RH. Amplatzer Duct Occluder device: a new technology for the closure of the moderate-to-large-sized patent ductus arteriosus. Expert Rev Med Devices. 2006 May;3(3):291-6. doi: 10.1586/17434440.3.3.291. PMID 16681450
- [Result] Moore JW, Levi DS, Moore SD, Schneider DJ, Berdjis F. Interventional treatment of patent ductus arteriosus in 2004. Catheter Cardiovasc Interv. 2005 Jan;64(1):91-101. doi: 10.1002/ccd.20243. PMID 15619281
- [Result] Perlo f, Joseph K.The Clinical Recognition of Congenital Heart Disease. Philadelphia: Saunders. Print.
- [Result] Gross RE, Hubbard JP. Landmark article Feb 25, 1939: Surgical ligation of a patent ductus arteriosus. Report of first successful case. By Robert E. Gross and John P. Hubbard. JAMA. 1984 Mar 2;251(9):1201-2. doi: 10.1001/jama.251.9.1201. No abstract available. PMID 6363741
- [Result] Kabra NS, Schmidt B, Roberts RS, Doyle LW, Papile L, Fanaroff A; Trial of Indomethacin Prophylaxis in Preterms Investigators. Neurosensory impairment after surgical closure of patent ductus arteriosus in extremely low birth weight infants: results from the Trial of Indomethacin Prophylaxis in Preterms. J Pediatr. 2007 Mar;150(3):229-34, 234.e1. doi: 10.1016/j.jpeds.2006.11.039. PMID 17307535
- [Result] Chorne N, Leonard C, Piecuch R, Clyman RI. Patent ductus arteriosus and its treatment as risk factors for neonatal and neurodevelopmental morbidity. Pediatrics. 2007 Jun;119(6):1165-74. doi: 10.1542/peds.2006-3124. PMID 17545385
- [Result] Teixeira LS, Shivananda SP, Stephens D, Van Arsdell G, McNamara PJ. Postoperative cardiorespiratory instability following ligation of the preterm ductus arteriosus is related to early need for intervention. J Perinatol. 2008 Dec;28(12):803-10. doi: 10.1038/jp.2008.101. Epub 2008 Jul 10. PMID 18615091
- [Result] Porstmann W, Wierny L, Warnke H, Gerstberger G, Romaniuk PA. Catheter closure of patent ductus arteriosus. 62 cases treated without thoracotomy. Radiol Clin North Am. 1971 Aug;9(2):203-18. No abstract available. PMID 4938290
- [Result] Weisz DE, McNamara PJ. Patent ductus arteriosus ligation and adverse outcomes: causality or bias? J Clin Neonatol. 2014 Apr;3(2):67-75. doi: 10.4103/2249-4847.134670. PMID 25024972
- [Result] Gruenstein DH, Ebeid M, Radtke W, Moore P, Holzer R, Justino H. Transcatheter closure of patent ductus arteriosus using the AMPLATZER duct occluder II (ADO II). Catheter Cardiovasc Interv. 2017 May;89(6):1118-1128. doi: 10.1002/ccd.26968. Epub 2017 Mar 4. PMID 28258658
- [Result] Kenny D, Morgan GJ, Bentham JR, Wilson N, Martin R, Tometzki A, Oslizlok P, Walsh KP. Early clinical experience with a modified Amplatzer ductal occluder for transcatheter arterial duct occlusion in infants and small children. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):534-40. doi: 10.1002/ccd.24522. Epub 2013 Jun 29. PMID 22718329
- [Result] Sungur M, Karakurt C, Ozbarlas N, Baspinar O. Closure of patent ductus arteriosus in children, small infants, and premature babies with Amplatzer duct occluder II additional sizes: multicenter study. Catheter Cardiovasc Interv. 2013 Aug 1;82(2):245-52. doi: 10.1002/ccd.24905. Epub 2013 Apr 8. PMID 23460349
- [Result] Bruckheimer E, Godfrey M, Dagan T, Levinzon M, Amir G, Birk E. The Amplatzer Duct Occluder II Additional Sizes device for transcatheter PDA closure: initial experience. Catheter Cardiovasc Interv. 2014 Jun 1;83(7):1097-101. doi: 10.1002/ccd.25445. Epub 2014 Mar 4. PMID 24532416
- [Result] Baspinar O, Sahin DA, Sulu A, Irdem A, Gokaslan G, Sivasli E, Kilinc M. Transcatheter closure of patent ductus arteriosus in under 6 kg and premature infants. J Interv Cardiol. 2015 Apr;28(2):180-9. doi: 10.1111/joic.12196. Epub 2015 Apr 2. PMID 25832591

DOCUMENTS (1):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04205877/Prot_000.pdf